CLINICAL TRIAL: NCT06125353
Title: The Effect of Melatonin Supplementation on Fatigue Symptoms During Chemotherapy Treatment of Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harokopio University (Other)
Responsible Party: Principal Investigator, Frantzeska Nimee, Principal Investigator, Harokopio University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 01052022; D231052019 (Other: The Ethics Committee of "IASO Hospital")
Record Dates: First submitted 2023-10-10; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Active Comparator): Participants in the Intervention group consumed one melatonin tablet per day, containing 1mg of melatonin, for a total of three months.
  Interventions: Dietary Supplement: Melatonin
- placebo group (No Intervention): Participants in this group were instructed to consume one placebo tablet (with water) every day for a total of three months. Melatonin and placebo tablets were of similar physical and sensory properties.

INTERVENTIONS:
Dietary Supplement: Melatonin — Patients of the Intervention group (melatonin group) received a personalized dietary plan based on the Mediterranean Diet, together with a booklet of lifestyle guidelines (nutritional and physical activity), all generated by a Clinical Decision Support System (CDSS). Moreover, participants in the Intervention group consumed one melatonin tablet per day, containing 1 mg of melatonin, together with water for a total of three months.
  Arms: intervention group

SUMMARY:
The aim of the present 3-month randomized, placebo-controlled trial was to evaluate whether adherence to Mediterranean Diet (MD) together with melatonin oral treatment or plaebo, would ameliorate Cancer Related Fatigue in Breast Cancer patients receiving chemotherapy treatment.

DETAILED DESCRIPTION:
Cancer related fatigue (CRF) is a common distressing complaint in breast cancer (BC) patients treated with chemotherapy. Nutrition quality plays a pivotal role in CRF, while an increased interest towards new pharmacological agents has been observed.

Melatonin, an endogenous hormone that regulates the human sleep-wake cycle, could alleviate CRF.

In the present randomized, placebo-controlled 3-month trial, we investigated the effects of melatonin intake (i.e., 1 mg/day) vs. placebo on CRF of BC patients. Melatonin and placebo tablets were of similar physical and sensory properties. In both arms, Mediterranean diet (MD) was implemented. Medical history, anthropometry and blood withdrawal were performed. CRF was evaluated by the Functional Assessment of Chronic Illness Therapy - Fatigue questionnaire and MD adherence by the MedDiet Score.

ELIGIBILITY:
Inclusion criteria:

1. adult women (≥ 18 years of age) with BC diagnosis who underwent chemotherapy at the time of invitation,
2. women receiving pharmacological treatment that did not interact with melatonin,
3. women receiving standard pharmacological treatment for at least last two months prior to study initiation,
4. patients with good performance status, as indicated by scoring "0 or 1" of the Eastern Cooperative Oncology Performance Status (ECOG PS) questionnaire [26],
5. patients not needing a transfusion, as indicated by hemoglobin ≥ 9 g/dL,
6. patients having the ability to understand and give a written statement of consent.

   Patients were excluded from the study when:
7. fatigue was attributed to conditions other than cancer e.g., uncontrolled hypothyroidism, hypercalcemia, congestive heart failure, chronic obstructive pulmonary disease,
8. using pharmacological agents for CRF or sleeping disorders prior to the study,
9. pharmacological treatment that was modified during the study or that could interact with melatonin,
10. diagnosed with gastrointestinal diseases that could affect absorption of nutrients such as inflammatory bowel diseases infections.
11. diagnosed with psychiatric disorders such as depression, psychosis, bipolar disorder, and receiving equivalent medication.
12. excessive alcohol consumption.
13. a lifestyle that can affect sleep patterns (e.g., night shifts).
14. patients with a poor clinical state as indicated by laboratory markers: creatinine clearance < 30 mL/min; aspartate aminotransferase (AST) > 3 x upper limit of normal (ULN); alanine aminotransferase (ALT) > 3 x ULN; bilirubin > 1 x ULN.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 56 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Cancer Related Fatigue | three months
  Whether melatonin can ameliorate cancer related fatigue in breast cancer patients. Cancer related fatigue was evaluated by the Functional Assessment of Chronic Illness Therapy - Fatigue questionnaire. It is a 40-item scale that assesses self-reported fatigue in terms of daily activities and function. It has five subscale domains: Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, Functional Well-Being, and Fatigue. For each question there are five answers (Not at all, A little bit, Somewhat, Quite a bit, Very much). Scoring ranges between 0 and 160. The higher the score, the better the participant's well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Skouroliakou, Dr, Study Director — Harokopio University
Locations (1):
- Iaso Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol